CLINICAL TRIAL: NCT00553033
Title: Prospective Evaluation of Laparoscopic Liver Resection
Brief Title: Laparoscopic Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Other Study IDs: LPSLIVER1
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Tumors
Keywords: Patients must be candidable to liver resection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- A
  Interventions: Procedure: Laparoscopic liver surgery

INTERVENTIONS:
Procedure: Laparoscopic liver surgery — Ultrasonic dissector, harmonic scalpel

SUMMARY:
The aim of this study is to evaluate the feasibility and safety of laparoscopic liver surgery.

DETAILED DESCRIPTION:
Perioperative course of patients undergoing liver resection is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* benign or malignant tumors
* tumor size less than 12 cm

Exclusion Criteria:

* Operations that required laparotomic procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients udergoing liver resection for benign or malignant tumors
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative Morbidity and mortality | Perioperative

SECONDARY OUTCOMES:
Patient satisfation | Perioperative
Patients satisfaction | Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Luca Aldrighetti, M.D PhD, Study Director — Department of Surgery - Liver Unit, Scientific Institute San Raffaele
Locations (1):
- Department of Surgery - Liver Unit, Scientific Institute San Raffaele, Milan, Milan, Italy

REFERENCES:
- [Result] Aldrighetti L, Pulitano C, Catena M, Arru M, Guzzetti E, Casati M, Comotti L, Ferla G. A prospective evaluation of laparoscopic versus open left lateral hepatic sectionectomy. J Gastrointest Surg. 2008 Mar;12(3):457-62. doi: 10.1007/s11605-007-0244-6. Epub 2007 Aug 14. PMID 17701265